CLINICAL TRIAL: NCT05044819
Title: A Long-term Safety Study to Assess the Potential for Chronic Liver Injury in Participants Treated With Epidiolex (Cannabidiol) Oral Solution
Brief Title: Assessment of Potential for Chronic Liver Injury in Participants Treated With Epidiolex (Cannabidiol) Oral Solution
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Jazz Pharmaceuticals Research UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWEP19022
Record Dates: First submitted 2021-08-30; First posted 2021-09-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Lennox Gastaut Syndrome; Dravet Syndrome; Tuberous Sclerosis Complex
Keywords: Liver injury; Liver fibrosis; Epidiolex; Cannabidiol
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsies, Myoclonic; Tuberous Sclerosis; Liver Cirrhosis | interventions — Cannabidiol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabidiol (Experimental): Cannabidiol solution 100 milligrams per milliliter (mg/mL) will be administered orally at a dose level of 5 mg/kg/day for 1 week, then increase to 10 mg/kg/day by the participant or their caregiver twice each day (morning and evening).
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Oral Cannabidiol solution 100 mg/mL
  Other Names: Epidiolex

SUMMARY:
This study will monitor for potential chronic liver injury and liver fibrosis, in participants treated with cannabidiol oral solution.

ELIGIBILITY:
Inclusion Criteria:

* Participant is within the approved age range as per labeling recommendations. Participants aged 1 to 3 years who are in the FibroScan subset will not undergo FibroScan assessments until they reach 4 years of age.
* Participant is either on existing Epidiolex therapy for treatment of a seizure disorder or is to be started on Epidiolex for treatment of an Food and Drug Administration (FDA)-approved indication.
* Participant is willing to refrain from strenuous exercise 48 to 72 hours prior to all study visits with the exception of unscheduled visits.
* Any non-pharmacological therapies (e.g., ketogenic diet) must also be stable up to 4 weeks prior to Screening Visit and expected to be stable throughout the duration of the study.

Exclusion Criteria:

* Participant is currently using or within 3 months of screening has used recreational or medicinal cannabis, or synthetic cannabinoid-based medications, not including Epidiolex if currently prescribed.
* Participant is not planning to abstain from using recreational cannabinoids or medicinal cannabis, or synthetic cannabinoid-based medications during the study.
* Female participant is pregnant (positive pregnancy test), lactating or planning pregnancy during the course of the study and for 3 months thereafter.
* Participant has any other significant disease or disorder which, in the opinion of the investigator, may either put the participant, other participants, or site staff at risk because of participation in the study, may influence the result of the study, or may affect the participant's ability to take part in the study
* Participant has diseases or disorders which are associated with liver fibrosis with a FibroScan score of ≥ 6.5 Kilopascals (where FibroScan results are available).
* Positive serology panel (including hepatitis B surface antigen and hepatitis C virus antibody) and/or positive human immunodeficiency virus antibody/p24 antigen screens at screening.
* Following a physical examination, if the participant has any abnormalities that, in the opinion of the investigator, would prevent the participant from safe participation in the study.
* Participant has significantly impaired hepatic function at Screening Visit alanine aminotransferase or aminotransferase > 3 x upper limit of normal (ULN), and total bilirubin > 2 x ULN or international normalized ratio > 1.5.
* Participant is planning to have epilepsy surgery or other major surgery within five years.
* Participant has or plans to have any medical device implanted that is contraindicated for use with FibroScan (only applicable for FibroScan subset), with the investigator consulting with the Sponsor as needed.
* Participation in any clinical trial involving an investigational medicinal product within 3 months prior to the Screening Visit or at any point during this study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Liver Fibrosis and Evaluable Fibrotic Changes as Determined and Assessed by an Independent Adjudication Committee | Screening, Day 365, Day 730, Day 1095, Day 1460, and Day 1825

SECONDARY OUTCOMES:
Change From Baseline in Aspartate Aminotransferase (AST) to Platelet Ratio Index | Baseline, Day 365, Day 730, Day 1095, Day 1460, and Day 1825
Change from Baseline in the Enhanced Liver Fibrosis Score | Baseline, Day 365, Day 730, Day 1095, Day 1460, and Day 1825
Change From Baseline in Fibrosis-4 | Baseline, Day 365, Day 730, Day 1095, Day 1460, and Day 1825
Change From Baseline in FibroScan Scoring (FibroScan subset only) | Baseline, Day 365, Day 730, Day 1095, Day 1460, and Day 1825
Number of Participants With Potential Drug-Induced Liver Injury (DILI) | Day 1, Day 365, Day 730, Day 1095, Day 1460, and Day 1825
Number of Participants with Severe Treatment-emergent Adverse Events (TEAEs) | Day 1, Day 365, Day 730, Day 1095, Day 1460, and Day 1825
Number of Participants With Clinically Significant Clinical Laboratory Findings | Day 1, Day 365, Day 730, Day 1095, Day 1460, and Day 1825
Number of Participants With Clinically Significant Physical Examinations | Day 1, Day 365, Day 730, Day 1095, Day 1460, and Day 1825

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Clinical Trial Site, Little Rock, Arkansas
  - Clinical Trial Site, Downey, California
  - Clinical Trial Site, Long Beach, California
  - Clinical Trial Site, Sacramento, California
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Augusta, Georgia
  - Clinical Trial Site, Wichita, Kansas
  - Clinical Trial Site, Lexington, Kentucky
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, New Brunswick, New Jersey
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Charlotte, North Carolina
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Oklahoma City, Oklahoma
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Charleston, South Carolina
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Round Rock, Texas
  - Clinical Trial Site, Winchester, Virginia

IPD SHARING:
Plan to Share IPD: No